CLINICAL TRIAL: NCT03404024
Title: A Phase II, Multicenter, Adaptive-design Study to Assess the Safety and Efficacy of VM202RY Injected Via Percutaneous Transendocardial Route in Subjects With Acute Myocardial Infarction
Brief Title: Safety and Efficacy Study of Gene Therapy for Acute Myocardial Infarction in Korea
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decided not to move forward with this study.
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMCAD-002
Record Dates: First submitted 2017-08-16; First posted 2018-01-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Heart Disease; Acute Myocardial Infarction
Keywords: gene therapy
MeSH Terms: conditions — Myocardial Ischemia | interventions — Hepatocyte Growth Factor; Sodium Chloride; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Stage 1-Low dose VM202RY (Experimental): Patients in this group will receive total 1mg of VM202RY. (4 sites of 0.25mg/0.5 mL VM202RY)
  Interventions: Biological: Stage 1-Low dose VM202RY; Device: C-Cathez® Catheter
- Stage 1-Middle dose VM202RY (Experimental): Patients in this group will receive total 2mg of VM202RY. (8 sites of 0.25mg/0.5 mL VM202RY)
  Interventions: Biological: Stage 1-Middle dose VM202RY; Device: C-Cathez® Catheter
- Stage 1-High dose VM202RY (Experimental): Patients in this group will receive total 3mg of VM202RY. (12 sites of 0.25mg/0.5 mL VM202RY)
  Interventions: Biological: Stage 1-High dose VM202RY; Device: C-Cathez® Catheter
- Stage 2-Placebo (Placebo Comparator): Patients in this group will receive 6mL of VM202RY vehicle. (12 sites of 0.5mL 0.9% NaCl, 1.1% sucrose)
  Interventions: Drug: Stage 2-Placebo; Device: C-Cathez® Catheter
- Stage 2-Low dose VM202RY (Experimental): Patients in this group will receive total 6mL of VM202RY and VM202RY vehicle. (The dose of VM202RY can be one of the three candidate-0.5mg VM202RY/1mg VM202RY/1.5mg VM202RY based on the tolerated dose result from Stage 1.)
  Interventions: Biological: Stage 2-Low dose VM202RY; Device: C-Cathez® Catheter
- Stage 2-High dose VM202RY (Experimental): Patients in this group will receive total 6mL of VM202RY and VM202RY vehicle. (The dose of VM202RY can be one of the three candidate-1mg VM202RY/2mg VM202RY/3mg VM202RY based on the tolerated dose result from Stage 1.)
  Interventions: Biological: Stage 2-High dose VM202RY; Device: C-Cathez® Catheter

INTERVENTIONS:
Biological: Stage 1-Low dose VM202RY — Day 0: 1mg of VM202RY (4 sites of 0.25mg/0.5mL VM202RY)
  Other Names: DNA Plasmid; Hepatocyte growth factor (HGF)-X7
  Arms: Stage 1-Low dose VM202RY
Biological: Stage 1-Middle dose VM202RY — Day 0: 2mg of VM202RY (8 sites of 0.25mg/0.5mL VM202RY)
  Other Names: DNA Plasmid; HGF-X7
  Arms: Stage 1-Middle dose VM202RY
Biological: Stage 1-High dose VM202RY — Day 0: 3mg of VM202RY (12 sites of 0.25mg/0.5mL VM202RY)
  Other Names: DNA Plasmid; HGF-X7
  Arms: Stage 1-High dose VM202RY
Drug: Stage 2-Placebo — Day 0: 6mL of VM202RY vehicle (12 sites of 0.5mL 1.1% sucrose/0.9% NaCl)
  Other Names: VM202RY vehicle; Sodium chloride, sucrose
  Arms: Stage 2-Placebo
Biological: Stage 2-Low dose VM202RY — Day 0: 6mL of VM202RY and VM202RY vehicle (total 12 site injections, low dose candidate-0.5mg VM202RY, 1mg VM202RY, 1.5mg VM202RY)
  Other Names: DNA plasmid; HGF-X7
  Arms: Stage 2-Low dose VM202RY
Biological: Stage 2-High dose VM202RY — Day 0: 6mL of VM202RY and VM202RY vehicle (total 12 site injections, high dose candidate-1mg VM202RY, 2mg VM202RY, 3mg VM202RY)
  Other Names: DNA Plasmid; HGF-X7
  Arms: Stage 2-High dose VM202RY
Device: C-Cathez® Catheter — Day 0 (Stage 1-Low dose VM202RY): 1mg of VM202RY (4 sites of 0.25mg/0.5mL VM202RY) Day 0 (Stage 1-Middle dose VM202RY): 2mg of VM202RY (8 sites of 0.25mg/0.5mL VM202RY) Day 0 (Stage 1-High dose VM202RY): 3mg of VM202RY (12 sites of 0.25mg/0.5mL VM202RY) Day 0 (Stage 2-Placebo): 6mL of VM202RY vehicle (12 sites of 0.5mL 1.1% sucrose/0.9% NaCl) Day 0 (Stage 2-Low dose VM202RY): 6mL of VM202RY and VM202RY vehicle (total 12 site injections, low dose candidate-0.5mg VM202RY, 1mg VM202RY, 1.5mg VM202RY) Day 0 (Stage 2-High dose VM202RY): 6mL of VM202RY and VM202RY vehicle (total 12 site injections, high dose candidate-1mg VM202RY, 2mg VM202RY, 3mg VM202RY)

SUMMARY:
The purpose of this study is to evaluate the safety and clinical efficacy of VM202RY injected via transendocardial route using C-Cathez® catheter (Celyad, S.A., Belgium) in subjects with AMI.

* Stage 1: Evaluation of safety and tolerability of VM202RY injection
* Stage 2: Evaluation of safety and efficacy of VM202RY injection

DETAILED DESCRIPTION:
Ischemic heart disease, a condition in which narrowed or blocked coronary arteries lead to ischemia in myocardium, is a group of disease that include: angina and myocardial infarction.

Acute myocardial infarction (AMI) predicts rapid progression of necrosis. AMI is a serious health condition that it's mortality rate is about 30% and also more likely to have a higher incidence of cardiac dysrhythmia or ventricular aneurysm.

Therapeutic angiogenesis is promising approach for the treatment of cardiovascular disease. 66 to 75% of coronary artery disease patients have insufficient coronary collaterals and 30% of myocardial infarction patients display inadequate myocardial perfusion although there are procedures like percutaneous coronary intervention or coronary artery bypass graft surgery.

In phase I study for ischemic heart disease, VM202RY appeared to have improved regional myocardial perfusion and wall thickness of the diastolic and systolic phases in the injected region. These results suggest that VM202RY improves the myocardial perfusion and inhibits cardiac remodeling in ischemic heart disease patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years to ≤ 75 years
2. Patients who underwent percutaneous coronary intervention (PCI) for the anterior wall infarction of left ventricle and had the elapsed time of 30 ± 2 days from the PCI, regardless of success or failure of myocardial revascularization in the anterior wall
3. Patients with > 20% to ≤ 45% of left ventricular ejection fraction via trans-thoracic echocardiography within 7 days prior to the study drug or placebo injection
4. Left ventricular wall thickness ≥ 8 mm via trans-thoracic echocardiography (however, the subject shall be included if 50% or greater of the left ventricular anterior wall is ≥8mm or injection site other than the left ventricular anterior wall is ≥ 8mm.)
5. If female of childbearing potential, negative urine pregnancy test at screening and using acceptable method of birth control during the study; if male, using barrier method of birth control during study
6. Be capable of understanding and complying with the protocol and signing the informed consent document prior to being subjected to any study related procedures.

Exclusion Criteria:

1. Severe systolic heart failure, NYHA Class III or IV
2. New York Heart Association (NYHA) functional class IV
3. History of recurrent ventricular tachycardia or cariogenic shock following PCI
4. Stroke or transient ischemic attack (TIA) within 180 days
5. Uncontrolled hypertension defined as systolic blood pressure ≥ 180 mmHg or diastolic ≥ 110 mmHg at screening and/or on the day of study drug or placebo injection
6. Sustained ventricular tachyarrhythmia or recurrent ventricular tachycardia
7. Implantation of automatic implantable cardioverter defibrillator (AICD)
8. On extracorporeal membrane oxygenator (ECMO)
9. History of ventricular fibrillation after PCI
10. Permanent pacemaker implantation (temporary pacemaker may be enrolled)
11. Subjects with aortic stenosis of moderate or greater degree, or with prosthetic aortic valve who may not be appropriate to use the C-CATHez® catheter due to the risk of injury during the interventional procedure through the valve
12. Atherosclerotic or other disease of the aorto-iliac system that would impede the safe passage of the C-CATHez®
13. Subjects with any serious comorbidities that the investigators deemed to be inappropriate to be enrolled
14. Patients with a recent history (< 5 years) of, or new screening finding of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence); patients with family history of colon cancer in any first degree relative are excluded unless they have undergone a colonoscopy in the last 12 months with negative findings
15. Elevated prostate-specific antigen (PSA) despite not having prostate cancer history
16. Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that preclude standard ophthalmologic examination Diagnosis of proliferative retinopathy or conditions that preclude standard ophthalmologic examination
17. Subjects currently receiving immunosuppressive medications, chemotherapy, or radiation therapy
18. Active infectious disease and/or positive Human Immunodeficiency Virus (HIV) or Human T-Cell lymphotropic viruses (HTLV) at screening
19. Active Hepatitis B or C infection as determined by Hepatitis B surface antibody (HBsAb), Hepatitis B core antibody (Immunoglobulin G and Immunoglobulin M; HBcAb), Hepatitis B surface antigen (HBsAg) and Hepatitis C antibodies (Anti-HCV) at screening
20. Specific laboratory values at screening including

    * Hemoglobin ≤ 9.0 g/dL, white blood cell (WBC) < 3,000 cells/μl, platelet count < 75,000/mm3
    * Creatinine > 2.0 mg/dL
    * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN)
    * Any other clinically significant lab abnormality which in the opinion of the investigator should be exclusionary
21. Subjects requiring > 100 mg daily of acetylsalicylic acid (ASA); subjects may be enrolled if willing/able to switch to ≤ 100 mg daily of ASA or to another medication
22. Subjects regularly taking cyclooxygenase (COX)-2 inhibiting drug(s) or non-specific COX-1/COX-2 inhibiting drugs, or high dose steroids (except inhaled steroids); subjects may be enrolled if willing/able to undergo medication wash-out prior to the first dosing and to refrain from taking these drugs for the duration of the study, and also if the subject is temporarily taking NSAID (non-steroidal anti-inflammatory drug) temporarily (≤ 7 days)
23. Patients that have undergone enhanced external pulsation (EECP) treatment within the last 6 months
24. Pregnancy or lactation
25. Severe comorbidity associated with a reduction of life expectancy of less than 1 year
26. Exposure to any previous experimental angiogenic therapy and/or myocardial laser therapy; or therapy with another investigational drug within 180 days of enrollment or participation in any concurrent study that may confound the results of this study
27. Major psychiatric disorder in the past 6 months
28. Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate
29. Deemed to be in unsuitable condition by the study investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-25 (Estimated); Primary Completion 2019-08-20 (Estimated); Study Completion 2019-08-20 (Estimated)

PRIMARY OUTCOMES:
Stage 1: MTD (maximum tolerated dose) | 6 months
  • MTD is defined as the dose level below the dose at which ≥ 33% of participants experienced DLT (dose limiting toxicity). The DLT assessment will be conducted on day 14. Toxicities more severe than grade 3 on the WHO toxicity scale will be designated as DLT. The dose where severe adverse events occur according to the Spilker classification will also be designated as DLT. The assessment will be conducted from the lowest dose to higher doses incrementally. MTD will be measured in milligrams (mg).
Stage 2: LVEF (left ventricular ejection fraction) measured by cardiac MRI | 6 months
  • The change in LVEF measured by cardiac MRI in VM202RY and placebo will be compared at 6 months after the treatment of VM202RY or Placebo by transendocardial injections using C-CATHez® catheter. LVEF will be measured in percentage (%).

SECONDARY OUTCOMES:
Change in left ventricular diameter (cardiac MRI) | 3 and 6 months
  The change in diameter of left ventricle will be measured in millimeters (mm), at months 3 and 6 using cardiac MRI.
Change in left ventricular diameter (TTE) | 3 and 6 months
  The change in diameter of left ventricle will be measured in millimeters (mm), at months 3 and 6 using TTE (transthoracic echocardiogram).
Change in left ventricular volume (cardiac MRI) | 3 and 6 months
  The change in volume of left ventricle will be measured in milliliters (mL), at months 3 and 6 using cardiac MRI.
Change in left ventricular volume (TTE) | 3 and 6 months
  The change in volume of left ventricle will be measured in milliliters (mL), at months 3 and 6 using TTE.
Change in cardiac output (cardiac MRI) | 3 and 6 months
  The change in cardiac output will be measured in liters per minute (L/min), at months 3 and 6 using cardiac MRI.
Change in cardiac output (TTE) | 3 and 6 months
  The change in cardiac output will be measured in liters per minute (L/min), at months 3 and 6 using TTE.
Change in LVEF (cardiac MRI) | 3 and 6 months
  The change in left ventricular ejection fraction will be measured in percentage (%), at months 3 and 6 using cardiac MRI.
Change in LVEF (TTE) | 3 and 6 months
  The change in left ventricular ejection fraction will be measured in percentage (%), at months 3 and 6 using TTE.
Change in wall motion score index (cardiac MRI) | 3 and 6 months
  The wall motion score index will be measured at months 3 and 6 using cardiac MRI.
Change in wall motion score index (TTE) | 3 and 6 months
  The wall motion score index will be measured at months 3 and 6 using TTE.
Change in myocardial wall thickness (cardiac MRI) | 3 and 6 months
  The change in myocardial wall thickness of the investigational-product or placebo injected area will be measured in millimeters (mm) at months 3 and 6 using cardiac MRI.
Change in extent of late enhancement of gadolinium (cardiac MRI) | 3 and 6 months
  The change in extent of late enhancement of gadolinium will be measured at months 3 and 6 using cardiac MRI.
Change in rest perfusion (cardiac MRI) | 3 and 6 months
  The change in rest perfusion will be measured in percentage (%) at months 3 and 6 using cardiac MRI.
Change in rest perfusion (myocardial SPECT) | 3 and 6 months
  The change in rest perfusion will be measured in percentage (%) at months 3 and 6 using myocardial SPECT.
Change in stress perfusion (cardiac MRI) | 3 and 6 months
  The change in stress perfusion will be measured in percentage (%) at months 3 and 6 using cardiac MRI.
Change in stress perfusion (myocardial SPECT) | 3 and 6 months
  The change in stress perfusion will be measured in percentage (%) at months 3 and 6 using myocardial SPECT.

CONTACTS AND LOCATIONS:
Overall Officials: Wook Bum Pyun, MD, PhD, Principal Investigator — Ewha Womans University
Locations (4):
- South Korea (4):
  - GangNeung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Ewha Womans University Medical Center, Seoul
  - KyungHee University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No